CLINICAL TRIAL: NCT05002374
Title: Application of Vestibular Rehabilitation Incorporated With Optokinetic Stimulation in Virtual Reality Environment in Patients With Peripheral Vestibular Dysfunction
Brief Title: Vestibular Rehabilitation Incorporated With Optokinetic Stimulation in Peripheral Vestibular Dysfunction Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Pei-Yun Lee, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-110-109
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Vestibular rehabilitation with optokinetic stimulation
- Control Group (Active Comparator)
  Interventions: Other: Vestibular rehabilitation

INTERVENTIONS:
Other: Vestibular rehabilitation with optokinetic stimulation — Vestibular rehabilitation incorporated with optokinetic stimulation in virtual reality environment for five consecutive days
  Arms: Experimental Group
Other: Vestibular rehabilitation — Customized vestibular rehabilitation for five consecutive days
  Arms: Control Group

SUMMARY:
Background Patients with peripheral vestibular dysfunction often complain of dizziness, blurred vision, imbalance and etc. Vestibular rehabilitation although has been proved to be an efficient method to improve the symptoms, the optimal treatment type, intensity and frequency is still unclear. Base on the mechanisms of vestibular rehabilitation, vestibular adaptation, substitution, and habituation, repeated practice and exposure to symptom-provoked movement could improve the symptoms. However, the symptom-provoked movement generated by only head and eye movement might not create sufficient threshold to induce vestibulo-ocular reflex adaptation. Practicing vestibular exercises in the same environment might be difficult for the patients to transfer learned ability to the real world environment. Therefore, optokinetic stimulation could potentially provide stronger visual-vestibular mismatch, and when combining with a virtual reality system could also simulate real world environment. Furthermore, an intensive training protocol on a daily basis might possibly promote the mechanisms of vestibular rehabilitation to enhance recovery from peripheral vestibular lesions. The purpose of this study is to investigate the efficacy of an intense vestibular rehabilitation programme incorporated with optokinetic stimulation in virtual reality environment on both subjective and objective symptoms in patients with peripheral vestibular dysfunction in the short and long term.

Methods This study will be an assessor-blind randomised controlled trial. Patients diagnosed as peripheral vestibular dysfunction aged between 20-80 years will be recruited and randomly allocated into two groups: vestibular rehabilitation incorporated with optokinetic stimulation in virtual reality (Group OKN) and vestibular rehabilitation only (Group C). Group C will receive customised vestibular rehabilitation, while Group OKN will receive the same exercise programme as Group C plus optokinetic stimulation provided in virtual environment. Both groups will receive vestibular rehabilitation intensively for five consecutive days with a trained physiotherapist, following with daily home exercise for two months. Self-perceived symptoms, spatial orientation, postural control and gait performance will be assessed prior to treatment (baseline), at the end of the five-day treatment, at four and eight weeks following the five-day training.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as peripheral vestibular dysfunction with bithermal caloric irrigation
* having one or more of the following subjective complains for longer than four weeks: vertigo/dizziness, disequilibrium, gait instability or motion sensitivity

Exclusion Criteria:

* central nervous system involvement
* active or poorly controlled migraine (more than one severe migraine a month)
* fluctuating symptoms e.g. Meniere's disease
* active benign paroxysmal positional vertigo (BPPV)
* have previous vestibular rehabilitation
* inability to attend sessions
* other medical conditions in the acute phase e.g. orthopaedic injury

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Subjective visual vertical test | Before treatment
  This test is to assess a person's perception of verticality. In this test, the subject is instructed to align a tilted illuminated line to self-perceived verticality in a completely darkened room. Differences between the subject's adjusted orientation and true spatial vertical are calculated as the subjective visual vertical.
Subjective visual vertical test | After the 5-day treatment
  This test is to assess a person's perception of verticality. In this test, the subject is instructed to align a tilted illuminated line to self-perceived verticality in a completely darkened room. Differences between the subject's adjusted orientation and true spatial vertical are calculated as the subjective visual vertical.
Subjective visual vertical test | At four weeks after the treatment
  This test is to assess a person's perception of verticality. In this test, the subject is instructed to align a tilted illuminated line to self-perceived verticality in a completely darkened room. Differences between the subject's adjusted orientation and true spatial vertical are calculated as the subjective visual vertical.
Subjective visual vertical test | At eight weeks after the treatment
  This test is to assess a person's perception of verticality. In this test, the subject is instructed to align a tilted illuminated line to self-perceived verticality in a completely darkened room. Differences between the subject's adjusted orientation and true spatial vertical are calculated as the subjective visual vertical.
Postural stability | Before treatment
  Standing postural stability under various conditions measured by a force platform
Postural stability | After the 5-day treatment
  Standing postural stability under various conditions measured by a force platform
Postural stability | At four weeks after the treatment
  Standing postural stability under various conditions measured by a force platform
Postural stability | At eight weeks after the treatment
  Standing postural stability under various conditions measured by a force platform

SECONDARY OUTCOMES:
The dizziness handicap inventory | Prior and after the 5-day treatment, and follow up at four and eight weeks after the treatment
  A 25-item self-report questionnaire assesses the impact of dizziness on daily life by measuring self-perceived handicap. The maximum score is 100. The higher the score, the more the perceived handicap due to dizziness.
The vestibular disorders activities of daily living scale | Prior and after the 5-day treatment, and follow up at four and eight weeks after the treatment
  This scale is used to assess the effects of vertigo and balance disorders on independence in everyday activities of daily living. This scale contains 28 items of self reporting questionnaire. It is divided into 3 subscales, which are functional, ambulation, and instrumental. The higher the score indicates higher dependence on the activities of daily living.
The hospital anxiety and depression scale | Prior and after the 5-day treatment, and follow up at four and eight weeks after the treatment
  This scale is used to assess depression and anxiety symptoms. It is a 14-item scale dividing into anxiety and depressive subscales. Scores of greater than or equal to 11 on either scale indicate a definitive case of anxiety or depression.
Gait performance | Prior and after the 5-day treatment, and follow up at four and eight weeks after the treatment
  Functional gait assessment, which is a 10-item gait assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yun Lee, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- Department of Physical Therapy, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No